CLINICAL TRIAL: NCT04540692
Title: NEOSAMBA Clinical Trial - Stage I
Brief Title: Evaluation of Sequencing of Anthracyclines and Taxanes for Locally Advanced HER2-negative Breast Cancer
Acronym: NEOSAMBA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Grupo Brasileiro de Estudos do Câncer de Mama (GBECAM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBECAM 0419; LACOG 0419 (Other: LACOG)
Record Dates: First submitted 2020-08-11; First posted 2020-09-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Paclitaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start with Cyclophosphamide + Doxorrubicin (Active Comparator): Patients will receive the following treatment schedule: Doxorubicin 60mg/m²; Cyclophosphamide 600mg/m² intravenously every 21 days for 3 cycles, followed by docetaxel 75-100mg/m2 intravenously every 21 days for 4 cycles or weekly paclitaxel 80mg/m2 for 12 weeks.
  Interventions: Drug: Cyclophosphamide + Doxorrubicin
- Start with Docetaxel or Paclitaxel (Experimental): Patients will receive the following treatment schedule: Docetaxel 75-100mg/m² intravenously every 21 days for 4 cycles or weekly paclitaxel 80mg/m² for 12 weeks, followed by Doxorubicin 60mg/m²; Cyclophosphamide 600mg/m² intravenously every 21 days, for 3 cycles.
  Interventions: Drug: Docetaxel or Paclitaxel

INTERVENTIONS:
Drug: Docetaxel or Paclitaxel — Treatment will start with Docetaxel 75-100mg/m² intravenously every 21 days for 4 cycles or weekly paclitaxel 80mg/m² for 12 weeks
  Other Names: Taxotere or Taxol
  Arms: Start with Docetaxel or Paclitaxel
Drug: Cyclophosphamide + Doxorrubicin — Treatment will start with Doxorubicin 60mg/m²; Cyclophosphamide 600mg/m² intravenously every 21 days for 3 cycles
  Other Names: Citoxan + Rubidox
  Arms: Start with Cyclophosphamide + Doxorrubicin

SUMMARY:
Phase III randomized clinical trial evaluating the sequencing of anthracyclines and taxanes in neoadjuvant therapy for locally advanced HER2-negative breast cancer.

DETAILED DESCRIPTION:
Multicenter, phase III, open-label, randomized clinical trial, which will include 494 patients randomized to two neoadjuvant chemotherapy arms. The treatment protocol will be the same in both groups, only the regimens sequences will be evaluated: starting with anthracycline versus taxane, with or without carboplatin for patients with triple negative subtype. The chemotherapy regimen will follow the institution's routine, which includes the use of CA in the anthracyclical phase and, in the taxane phase, the use of docetaxel every 21 days or weekly paclitaxel. The rest of the treatment (surgery, radiotherapy, hormone therapy) will not be part of the study and will be carried out according to institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, with at least 18 years old on the day of signing the free and informed consent;
* Invasive breast carcinoma stage III (RH positive) or IIB/III (RH negative), according to TNM 8th edition; Histologically confirmed diagnosis of invasive breast carcinoma (with any histology), HER-2 negative;
* The participant (or legally acceptable representative, if applicable) provides written informed consent for the study;
* The participant must agree to use a contraceptive as detailed in Appendix B of this protocol during the treatment period and for at least 120 days after the last dose of the study treatment;
* Have a functional capacity according to the Eastern Cooperative Oncology Group (ECOG) from 0 to 2. The evaluation of the ECOG must be carried out within 7 days before the inclusion date.
* Have adequate organic function. The samples must be collected within 60 days before the start of the study treatment;
* Have adequate cardiac function as assessed by echocardiogram or MUGA performed up to 60 days before the start of treatment under study.

Exclusion Criteria:

- Individuals who do not meet the inclusion criteria above-mentioned.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | An average of 8 years
  Defined as the time elapsed between the date of randomization and the date of invasive recurrence (excludes carcinoma in situ) or death, whichever comes first..

CONTACTS AND LOCATIONS:
Overall Officials: José Bines, Principal Investigator — Grupo Brasileiro de Estudos do Câncer de Mama (GBECAM)
Locations (18):
- Brazil (18):
  - Hospital Evangélico de Cachoeiro de Itapemirim - Centro de Pesquisas Clínicas em Oncologia (CPCO), Cachoeiro de Itapemirim, Espírito Santo
  - Santa Casa de Misericórdia da Bahia - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Centro de Pesquisa do Hospital Araújo Jorge, Goiânia, Goiás
  - ICTR - Instituto do Câncer e Transplante de Curitiba, Curitiba, Paraná
  - HUEM/CEON - Hospital Universitário Evangélico Mackenzie, Curitiba, Paraná
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - IMIP - Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Hospital Universitário Oswaldo Cruz (UNIPECLIN), Recife, Pernambuco
  - HINJA - Hospital Jardim Amália, Volta Redonda, Rio de Janeiro
  - HCPA - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncológicas, Florianópolis, Santa Catarina
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista (UPECLIN), Botucatu, São Paulo
  - Faculdade de Ciências Médicas da Unicamp, Campinas, São Paulo
  - Hospital de Amor Jales - Hospital de Câncer de Barretos, Jales, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - ICESP - Instituto do Câncer do Estado de São Paulo, São Paulo
  - IBCC Oncologia - Núcleo de Pesquisa São Camilo, São Paulo